CLINICAL TRIAL: NCT03220867
Title: A Single-Dose, Randomized, Open-Label, Two-Treatment, Two-Period, Two-Cohort, Crossover Study to Assess the Bioequivalence of Xian Risperdal Tablets Under Fasting and Fed Conditions in Chinese Healthy Subjects Compared With Gurabo Risperdal Tablets
Brief Title: Bioequivalence Study of Xian Risperdal Tablets Compared With Gurabo Risperdal Tablets Under Fasting and Fed Conditions in Chinese Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: CFDA announced Xi'An Risperdal as reference drug, no need for this BE trial from both scientific and ethical perspective.
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108341; R064766SCH1013 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence: AB (Experimental): Participants in cohort 1 (fasting) and cohort 2 (fed) will receive 1 milligram (mg) risperidone administered as Xian Risperdal (test) 1*1 mg oral tablet (Treatment A) on Day 1 in Period 1 followed by 1 mg risperidone administered as Gurabo Risperdal (reference) 1*1 mg oral tablet (Treatment B) on Day 1 in period 2. There will be a washout period of at least 10 days between treatments.
  Interventions: Drug: Risperidone: Xian Risperdal (test); Drug: Risperidone: Gurabo Risperdal (reference)
- Treatment Sequence: BA (Experimental): Participants in cohort 1 (fasting) and cohort 2 (fed) will receive Treatment B on Day 1 in period 1 followed by Treatment A on Day 1 in period 2. There will be a washout period of at least 10 days between treatments.
  Interventions: Drug: Risperidone: Xian Risperdal (test); Drug: Risperidone: Gurabo Risperdal (reference)

INTERVENTIONS:
Drug: Risperidone: Xian Risperdal (test) — Participants will receive 1*1 mg tablet of Xian Risperdal under fasting or fed condition.
  Other Names: JNJ-410397-AAA
Drug: Risperidone: Gurabo Risperdal (reference) — Participants will receive 1*1 mg tablet of Gurabo Risperdal under fasting or fed condition.

SUMMARY:
The primary purpose of this study is to assess the bioequivalence of Xian Risperdal compared with Gurabo Risperdal in Chinese healthy participants under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study and adhere to the prohibitions and restrictions specified in this protocol
* If a woman, must have a negative serum pregnancy test at screening and on Day -1 of each treatment period
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 2 months after receiving the last dose of study drug
* Body mass index (BMI), weight (kilogram [kg])/height^2 (meter [m]^2) between 19.0 and 28.0 kg/m^2, inclusive; body weight not less than 50 kg
* After being supine for 5 minutes, systolic blood pressure between 90 and 140 millimeter of mercury (mmHg), inclusive; diastolic blood pressure between 60 and 90 mmHg, inclusive; heart rate between 50 and 100 beats per minute (bpm), inclusive

Exclusion Criteria:

* Presence of orthostatic hypertension at screening, defined as a fall in systolic blood pressure of at least 20 mmHg or diastolic blood pressure of at least 10 mmHg compared to supine position when the participant assumes a standing position
* Positive test for drug screening, such as cannabinoids, opiates, cocaine, amphetamines, benzodiazepines, hallucinogens or barbiturates on Day -1 of each treatment period
* Drug abusers or use of soft drugs (example [eg], cannabis) within 3 months prior to the study or hard drugs (eg cocaine, benzene cyclohexylidene, etc.) within 1 year prior to the study
* Received an experimental drug or used an experimental medical device within 3 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Positive test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C antibodies or syphilis serum test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-04-27 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 15, 30, 45 minutes post-dose, and 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 48, 72 and 96 hours post-dose
  Maximum observed plasma concentration (Cmax) will be assessed.
Area Under Concentration-Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) | Pre-dose, 15, 30, 45 minutes post-dose, and 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 48, 72 and 96 hours post-dose
  Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Pre-dose, 15, 30, 45 minutes post-dose, and 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 48, 72 and 96 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant. AUC (0-infinity) will be assessed.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to approximately 29 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (1):
- Beijing Shijitan Hospital, Beijing, China